CLINICAL TRIAL: NCT01251068
Title: Measurement of Cerebral and Peripheric Tissue Oxygenation in Anemic Preterm Infants Who Underwent Blood Transfusion:A Near Infrared Spectroscopy Study.
Brief Title: Measurement of Cerebral and Peripheric Tissue Oxygenation in Anemic Preterm Infants Who Underwent Blood Transfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Neonatal Intensive Care Unit
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-11

CONDITIONS: Anemic Preterms, Cerebral Oxygenation,Somatic Oxygenation,Blood Transfusion
Keywords: anemic preterms, cerebral oxygenation,somatic oxygenation, blood transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gest age, cerebral ,somatic oxygenation measurement (Experimental)
  Interventions: Device: near infrared spectroscopy: invos 5100; Device: INVOS 5100; Device: near infrared spectroscopy device

INTERVENTIONS:
Device: near infrared spectroscopy: invos 5100 — duration:six hours
Device: INVOS 5100 — NIRS device used in this study, the optical field includes a volume of tissue approximately 2 cm deep to the surface probe with a 4-mm source-detector distance, and thus, organ-specific monitoring is feasible in small patients. With informed consent, we applied NIRS probes to the forehead and the lower extremity for cerebral (rSO2C) and peripheric (rSO2P) regional oxygen saturation measurements.
Device: near infrared spectroscopy device — NIRS device used in this study, the optical field includes a volume of tissue approximately 2 cm deep to the surface probe with a 4-mm source-detector distance, and thus, organ-specific monitoring is feasible in small patients. With informed consent, we applied NIRS probes to the forehead and the lower extremity for cerebral (rSO2C) and peripheric (rSO2P) regional oxygen saturation measurements.

SUMMARY:
Near infrared spectroscopy offers the possibility of noninvasive and continuous bedside investigation of cerebral oxygenation in newborn infants. Using this technique we investigated the relationship between changes in cerebral oxygenation and hemodynamics, and changes in some physiological variables during blood transfusion in anaemic preterm infants.

ELIGIBILITY:
Inclusion Criteria: <32 gestational age and/or <1500gr.,>30th day preterm infants -

Exclusion Criteria:sepsis,shock,severe intracranial hemorrhage,NEC,abdominal and cranial surgery

-

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Cerebral and peripheric oxygenation measurements in anemic preterm infants. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Maternity Teaching Hospital, Ankara, Hamamönü, Turkey (Türkiye)